CLINICAL TRIAL: NCT04698252
Title: Local Therapy for Hormone Receptor-positive Oligometastatic Breast Cancer - a Phase II Randomized Trial
Brief Title: Local Therapy for ER/PR-positive Oligometastatic Breast Cancer
Acronym: LARA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1752/20
Record Dates: First submitted 2020-12-04; First posted 2021-01-06 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Oligometastasis; Hormone Receptor Positive; Surgery; Radiotherapy; Radiofrequency ablation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic therapy (No Intervention): Patients will receive standard of care with systemic therapy alone.
- Local therapy + systemic therapy (Experimental): In addition to systemic therapy, patients will receive local therapy for all oligometastatic sites. Options of local therapy will be radiotherapy, radiofrequency ablation, and/ or surgery.
  Interventions: Radiation: Radiotherapy; Procedure: Surgery; Other: Radiofrequency ablation

INTERVENTIONS:
Radiation: Radiotherapy — Radiation therapy for oligometastatic sites
  Arms: Local therapy + systemic therapy
Procedure: Surgery — Surgery for oligometastatic sites
  Arms: Local therapy + systemic therapy
Other: Radiofrequency ablation — Radiofrequency ablation for oligometastatic sites
  Arms: Local therapy + systemic therapy

SUMMARY:
Randomized phase 2 trial to evaluate the efficacy of local therapy for oligometastasis from ER/PR-positive breast cancer. The study hypothesis is that local therapy in addition to systemic therapy improves progression-free survival in comparison with systemic therapy alone.

DETAILED DESCRIPTION:
Patients with estrogen receptor/ progesterone receptor-positive oligometastatic breast cancer with disease controlled after at least six months of systemic therapy will be enrolled in the study. Patients will be randomized to receive local therapy for oligometastatic sites in addition to systemic therapy or systemic therapy alone. Local therapy strategies will include surgery, radiotherapy, and radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* ≥ 18 years of age
* Histologically confirmed invasive breast cancer, with oligometastatic disease defined as one of the following criteria: 1) One to four bone lesions; 2) One to four lung and/ or hepatic lesions; 3) Distant metastasis limited to ipsilateral cervical lymph nodes; 4) Distant metastasis limited to contralateral axillary lymph nodes
* Oligometastatic sites amenable to treatment with a local therapy modality, including surgical resection, stereotactic radiotherapy, or radiofrequency ablation
* Estrogen receptor-positive and/ or progesterone receptor-positive breast cancer
* Partial response or stable disease after at least six months of systemic therapy for breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Measurable or non-measuble disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Life expectancy of at least 12 weeks
* For women in childbearing age, negative pregnancy test until 21 days before the date of study enrollment.
* Signed informed consent form
* Disposition and aptitude to fulfill the study protocol during the study duration

Exclusion Criteria:

* HER2-positive breast cancer
* Progressive disease during the last systemic treatment received for metastatic disease
* Previous local therapy for distant metastasis
* Current or previous history of severe diseases, such as clinically relevant heart failure, acute myocardium infarction in the last six months, chronic obstructive lung disease, HIV infection, chronic active hepatitis B or C infection, current serious uncontrolled infections or other severe diseases that may impact patients' expected survival)
* Current or previous history of other invasive malignancy within the last five years, excluding non-melanoma skin cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) | from baseline up to 2 years
  PFS will be defined as the time from randomization until the date of progression or death. 2-year PFS rate will represent the probability of a patient being free of progression after 2 years of randomization and will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall-survival (OS) | from baseline up to 10 years
  OS will be calculated from the date of randomization until the date of death from any cause.
Local therapy complication rate | from baseline up to 10 years
  Local therapy complications will be registered, including the occurrence of bleeding, local infections, pneumothorax, or other events attributed to local therapy by the medical team. Acute complications will be considered as those occurring until one month after procedure, while late complication will be those occurring later than one month.
1. European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30) | from baseline up to 1 year
  The EORTC QLQ-C30 provide points for questions related to global health status, functional scales, and symptom scales, providing scores ranging from 0-100. Higher scores represent higher health status, higher functioning, and higher symptom burden.
2. European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Breast Cancer (QLQ-BR23) | from baseline up to 1 year
  EORTC-QLQ-BR23 is composed of questions related to functional scales and symptom scales specific for breast cancer, providing scores ranging from 0-100. Higher scores for functional scales represent better functioning, while higher scores for symptom scales represent higher levels of symptoms.
Chemotherapy-free survival | from baseline up to 10 years
  Chemotherapy-free survival will be calculated from the date of randomization until the first date of application of a new chemotherapy line.
Subgroup analysis - PFS according to type of metastatic disease (de novo versus recurrent) and metastatic sites | from baseline up to 10 years
  PFS will be calculated for subgroups, according to type of metastatic disease (de novo versus recurrent) and sites of oligometastasis

CONTACTS AND LOCATIONS:
Overall Officials: Renata C. Bonadio, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil